CLINICAL TRIAL: NCT04606433
Title: An Open, Multicenter, Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics/Pharmacokinetics, and Antitumor Activity of GNC-038 Quad-specific Antibody Injection in Relapsed or Refractory Non-Hodgkin's Lymphoma, Relapsed or Refractory Acute Lymphoblastic Leukemia, and Refractory or Metastatic Solid Tumors
Brief Title: Phase I Clinical Study of GNC-038 in Patients With Non-Hodgkin's Lymphoma or Acute Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: SystImmune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GNC-038-101
Record Dates: First submitted 2020-10-08; First posted 2020-10-28 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Non Hodgkin Lymphoma; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): The patients received intravenous infusion of GNC-038 for 1 cycle. After the completion of 2 cycles of treatment, participants with no unbearable ae could proceed to the 3rd and 4th cycles of treatment. After four cycles of treatment, participants with clinical benefits could also receive four additional cycles of the same dose.
  Interventions: Drug: GNC-038

INTERVENTIONS:
Drug: GNC-038 — Administration by intravenous infusion.

SUMMARY:
An open, multicenter, Phase I clinical study to evaluate the safety, tolerability, pharmacokinetics/pharmacokinetics, and antitumor activity of GNC-038 quad-specific antibody injection in relapsed or refractory non-Hodgkin's lymphoma, relapsed or refractory acute lymphoblastic leukemia, and refractory or metastatic solid tumors.

DETAILED DESCRIPTION:
Phase Ia: To observe the safety and tolerability of GNC-038 in patients with relapsed or refractory non-Hodgkin lymphoma (R/R NHL)/relapsed or refractory acute lymphoblastic leukemia (R/R ALL), To determine the maximum tolerated dose (MTD) or maximum administration dose (MAD) and dose-limiting toxicity (DLT) of GNC-038 without MTD and recommend the dose for subsequent clinical studies. Phase Ib: To further observe the safety and tolerability of GNC-038 at the Phase Ia recommended dose to determine the Phase II recommended dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

1. The participants could understand and sign the informed consent form, and must participate voluntarily.
2. No gender limit.
3. Age: ≥18 years old.
4. Expected survival time ≥ 3 months.
5. Histologically or cytologically confirmed non-Hodgkin's lymphoma or acute lymphoblastic leukemia.
6. Patients with relapsed refractory non-Hodgkin lymphoma (R/R NHL). Specifically, patients who relapsed for the first time and still progressed during second-line treatment; Patients with relapse after second-line or multiline therapy; Refractory patients showed no remission or progress after full dose and full cycle use of standard or current clinically commonly selected combination therapy regimen, and no remission or progress after replacement of second-line regimen; Patients with relapsed or refractory non-Hodgkin lymphoma who were determined to have no or no other treatments available/intolerant.
7. Relapsed or refractory acute lymphoblastic leukemia (R/R ALL), including: no response after more than 6 weeks of induction chemotherapy, or no response after 2 cycles of induction chemotherapy; A second or more recurrence of bone marrow; Or relapse for the first time after chemotherapy with no remission after at least 1 cycle of salvage therapy; Bone marrow recurrence after autologous stem cell transplantation (auto-HSCT); Patients with relapsed or refractory acute lymphoblastic leukemia were determined to have no or no other treatments/intolerant.
8. Patients with Philadelphia chromosome positive (Ph+) ALL who are intolerant to or fail to treat 1 and/or 2 generation tyrosine kinase inhibitors (TKI), or Ph+ALL who have a T315I mutation, do not require TKI salvage therapy.
9. For patients with NHL, there were measurable lesions in the screening period (lymph node lesions with any length ≥1.5cm or exodal lesions with any length > 1.0cm); CLL/SLL: peripheral blood leukemia cells ≥5.0×109/L; Or lymph node lesions of any length ≥1.5cm; WM: IgM> 2 x ULN.
10. For AITL and NK/T lymphoma, a membrane CD3 negative test is required.
11. Physical status score ECOG ≤2 points.
12. The toxicity of previous antitumor therapy has returned to ≤ Class 1 as defined by NCI-CTCAE v5.0 (except for toxicities that the investigators judged to be of no safety risk, such as alopecia, grade 2 peripheral neurotoxicity, and stable hypothyroidism after hormone replacement therapy).
13. The organ function level meets the following requirements: Bone marrow function (for NHL patients only) : without blood transfusion within 7 days prior to screening, without G-CSF (without long-acting rising white needle within 2 weeks), and without drug correction: Absolute neutrophil count (ANC) ≥1.0×109/L (≥0.5×109/L for subjects with bone marrow infiltration); Hemoglobin ≥80 g/L (≥70g/L for subjects with bone marrow infiltration); Platelet count ≥50×109/L; Liver function: Total bilirubin ≤1.5 ULN (Gilbert's syndrome ≤3 ULN), transaminase (AST/ALT) ≤2.5ULN (in subjects with tumor invasive changes in the liver ≤5.0 ULN), and/or alkaline phosphatase ≤5 ULN when not corrected with hepatoprotective drugs within 7 days prior to screening; Renal function: creatinine (Cr) ≤1.5 ULN and creatinine clearance (Ccr) ≥50 ml/min (based on the center's calculation criteria). The investigators judged renal function intact without injury, except that abnormal creatinine index was caused by tumor. Coagulation function: fibrinogen ≥1.5g/L; Activated partial thromboplastin time (APTT) ≤1.5×ULN; Prothrombin time (PT) ≤1.5×ULN.
14. Fertile female subjects or male subjects with fertile partners must use highly effective contraception from 7 days before the first dose until 6 months after the last dose. A fertile female subject must have a negative serum pregnancy test within 7 days prior to initial dosing.
15. The subject is able and willing to comply with visits, treatment plans, laboratory tests, and other study-related procedures as specified in the study protocol.

Exclusion Criteria:

1. Live virus vaccine (including attenuated live vaccine) was administered within 28 days prior to administration in this study.
2. Patients who received major surgery within 28 days prior to administration of the drug or planned to undergo major surgery during the study period (except for procedures such as puncture or lymph node biopsy).
3. Defined as ≥ Grade 3 pulmonary diseases according to NCI-CTCAE v5.0; Patients with present or history of interstitial lung disease (ILD).
4. Systemic serious infections occurred within 1 week before screening, including but not limited to severe pneumonia caused by fungi, bacteria and viruses, bacteremia or serious infectious complications.
5. Active tuberculosis.
6. People with active autoimmune disease, or a history of autoimmune disease, Including but not limited to Crohn's disease, ulcerative colitis, systemic lupus erythematosus, sarcoidosis, Wegener syndrome, polyvasculitis granulomatosis, autoimmune hepatitis, systemic sclerosing disease, autoimmune vasculitis, autoimmune neuropathy (Guillain-Barre syndrome), etc. Exceptions include type I diabetes, hypothyroidism stable on hormone replacement therapy (including hypothyroidism caused by autoimmune thyroid disease), psoriasis or vitiligo that does not require systemic therapy, and B-cell autoimmune disease.
7. Non-melanoma skin cancer in situ, superficial bladder cancer in situ, cervical cancer in situ, gastrointestinal intramucosal cancer, breast cancer, localized prostate cancer and other malignant tumors that were combined with other malignant tumors within 5 years prior to the first administration of the drug, and those that had been cured and had not recurred within 5 years were excluded.
8. HBsAg positive; HBcAb positive and HBV-DNA detection ≥ lower limit of detection value; HCV antibody positive and HCV-RNA≥ lower limit of detection value; HIV antibody positive.
9. Poorly controlled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg).
10. A history of severe cardiovascular and cerebrovascular diseases, including but not limited to: severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, degree III atrioventricular block, etc.; At rest, the QT interval was prolonged (QTc > 450 msec in men or 470msec in women); Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events occurred within 6 months prior to initial administration; There is heart failure ≥II on the New York Heart Association (NYHA) cardiac function scale.
11. Patients with a history of allergy to recombinant humanized antibodies or to any excipient component of GNC-038.
12. Pregnant or breastfeeding women.
13. Patients with central nervous system invasion.
14. Previous recipients of organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT).
15. Autologous hematopoietic stem cell transplantation (AutoHSCT) was performed within 12 weeks prior to initiation of GNC-038 therapy.
16. Immunosuppressants are being used, including but not limited to: cyclosporine, tacrolimus, etc., within 2 weeks prior to treatment with GNC-038; GNC-038 received high doses of glucocorticoids within 2 weeks prior to treatment (longer than 14 days, daily steady dose > 30mg of prednisone or equal doses of other corticosteroids), except for patients with R/R ALL, Dexamethasone should be symptomatic when R/R ALL patients have more than 50% bone marrow protocells or peripheral protocells ≥15000/μL during the screening period (see 4.6.2 Availability of drugs during the trial).
17. Received radiotherapy within 4 weeks prior to initiation of GNC-038 treatment.
18. Patients with NHL who had received anti-CD20 or anti-CD79B therapy within 4 weeks before starting GNC-038 therapy continued to respond; ALL patients were treated with TKI, anti-CD19 or anti-CD22 within 4 weeks prior to GNC-038 and still responded, and were treated with bonatumab (CD19×CD3) and izumab - oxomicin (CD22-ADC) within 4 weeks prior to treatment.
19. Received chemotherapy and small-molecule targeted therapy within 2 weeks prior to treatment.
20. Received CAR T therapy within 12 weeks prior to initiation of GNC-038 therapy.
21. Participants in any other clinical trial within 4 weeks prior to administration of this trial.
22. Other conditions deemed unsuitable for participation in this clinical trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Up to 14 days after the first dose
  The incidence and severity of adverse events (TEAE) during treatment were graded according to the National Cancer Institute Standard for Common Terminology for Adverse Events (NCI-CTCAE, v5.0).
Maximum tolerated dose (MTD) or maximum administrated dose (MAD) | Up to 14 days after the first dose
  In the dose increment stage, the highest dose whose estimated DLT rate is closest to the target DLT rate but does not exceed the upper bound of the equivalent interval of DLT rate is selected as MTD.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of GNC-038. The type, frequency and severity of TEAE will be evaluated during the treatment of GNC-038.
The recommended dose for future clinical study | Up to 14 days after the first dose of GNC-038
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of GNC-038.

SECONDARY OUTCOMES:
Adverse Events of special interest (AESI) | Up to approximately 24 months
  AESI is an event of scientific and medical interest specific to the sponsor's product or research project.
Cmax: Maximum serum concentration of GNC-038 | Up to 14 days after the first dose of GNC-038
  Maximum serum concentration (Cmax) of GNC-038 will be investigated.
Css: Concentration of GNC-038 at steady state plateau | Up to 14 days after the first dose of GNC-038
  Concentration of GNC-038 at steady state plateau will be investigated.
Tmax: Time to maximum serum concentration (Tmax) of GNC-038 | Up to 14 days after the first dose of GNC-038
  Time to maximum serum concentration (Tmax) of GNC-038 will be investigated.
T1/2: Half-life of GNC-038 | Up to 14 days after the first dose of GNC-038
  Half-life (T1/2) of GNC-038 will be investigated.
AUC0-inf: Area under the serum concentration-time curve from time 0 to infinity | Up to 14 days after the first dose of GNC-038
  Blood concentration - Area under time line.
AUC0-t: Area under the serum concentration-time curve from time 0 to the time of the last measurable concentration | Up to 14 days after the first dose of GNC-038
  Blood concentration - Area under time line.
CL: Clearance in the serum of GNC-038 per unit of time | Up to 14 days after the first dose of GNC-038
  To study the serum clearance rate of GNC-038 per unit time.
Incidence and titer of ADA (Anti-drug antibody) | Up to approximately 24 months
  Frequency and titer of anti-GNC-038 antibody (ADA) will be evaluated.
Incidence and titer of Nab (Neutralizing antibody) | Up to approximately 24 months
  Incidence and titer of Nab of GNC-038 will be evaluated.
ORR (Objective Response Rate ) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
DCR (Disease Control Rate) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
PFS (Progression-free Survival) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of GNC-038 to the first date of either disease progression or death, whichever occurs first.
DOR (Duration of Response) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Principal Investigator — Hematology Hospital, Chinese Academy of Medical Sciences; Junyuan Qi, Principal Investigator — Hematology Hospital, Chinese Academy of Medical Sciences
Locations (10):
- China (10):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Shanghai Tongji Hospital, Shanghai, Shanghai Municipality
  - Hematology Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No